CLINICAL TRIAL: NCT06711458
Title: Using Generative Artificial Intelligence to Transform Discharge Summaries Into Patient-Friendly Language and Format
Brief Title: Using Generative Artificial Intelligence (AI) to Create Patient-Friendly Discharge Summaries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-01544
Record Dates: First submitted 2024-11-27; First posted 2024-12-02 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Hospital Discharge Summary Understanding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Generative AI Discharge Instructions (Experimental): At the time of discharge, patients will receive patient-friendly discharge instructions generated by GPT-4, an advanced natural language processing model, with the aim of enhancing patient readability and understandability in the discharge information.
  Interventions: Behavioral: AI-Generated Discharge Instructions
- Standard of Care Discharge Instructions (Active Comparator): At the time of discharge, patients will receive standard discharge instructions (i.e., not generated by GPT-4).
  Interventions: Behavioral: Standard of Care Discharge Instructions

INTERVENTIONS:
Behavioral: AI-Generated Discharge Instructions — Patient-friendly hospital discharge instructions generated by GPT-4, an advanced natural language processing model.
  Arms: Generative AI Discharge Instructions
Behavioral: Standard of Care Discharge Instructions — Standard hospital discharge instructions.
  Arms: Standard of Care Discharge Instructions

SUMMARY:
This will be an open-label, parallel-group, randomized trial. Patients will be randomized to review the patient-friendly discharge instructions at the time of discharge (intervention group) vs the standard of care. The intervention differs from the standard of care in that patients will be given additional medical documentation in the intervention group.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to Inpatient Medicine unit at NYULH
* Able to read and understand English
* Willing and able to consent to this research

Exclusion Criteria:

* Inpatient Hospice
* Discharged on home hospice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2025-01-29 (Actual); Primary Completion 2025-05-22 (Actual); Study Completion 2025-05-22 (Actual)

PRIMARY OUTCOMES:
Number of Summaries with Positive Outcome on Composite Measure of Readability and Understandability | Day 1 (At Discharge)
  This is a composite outcome measure. Readability of discharge summaries will be measured using the Flesch-Kincaid Grade Level assessment, which measures how challenging a text may be for readers. Scores on the Flesch-Kincaid assessment are rated as follows:
  0-3: Basic reading level, (kindergarten or elementary school) 3-6: Basic reading level, (elementary school ) 6-9: Average reading level, (middle school) 9-12: Average reading level, (high school) 11-18: Skilled readers.
  Understandability will be evaluated by the presence of simplified description of primary diagnosis and hospital intervention.
  Summaries with both 1) presence of simplified description of primary diagnosis and hospital intervention, and 2) a Flesch-Kincaid grade level greater than or equal to 6 and less than 8, will be considered to have a "positive outcome."

SECONDARY OUTCOMES:
Changes made to AI-Generated Content | Day 1 (At Discharge)
  Changes made to content will be assessed using edit distance.
AI-Generated Content Perception Survey: Safety | Day 1 (At Discharge)
  Patients will be given a survey in which they are asked whether they feel safe with the discharge instructions they were provided. The total score is the number of participants who respond "Yes, definitely" or "Yes, somewhat" to the question.
AI-Generated Content Perception Survey: Understandability | Day 1 (At Discharge)
  Patients will be given a survey in which they are asked whether the instructions were easy to understand. The total score is the number of participants who respond "Yes, definitely" or "Yes, somewhat" to the question.
AI-Generated Content Perception Survey: Empathy | Day 1 (At Discharge)
  Patients will be given a survey in which they are asked whether the instructions were written in an empathetic manner. The total score is the number of participants who respond "Yes, definitely" or "Yes, somewhat" to the question.

CONTACTS AND LOCATIONS:
Overall Officials: Jonah Zaretsky, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Data collected from usual clinical care; these data cannot be easily deidentified or shared.